CLINICAL TRIAL: NCT04075370
Title: Exploring Compensation to Maintain Cognitive Function in Adults Newly Diagnosed With Brain Cancer
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00092580
Record Dates: First submitted 2019-08-26; First posted 2019-08-30 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Primary Brain Tumor; Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for biomarker testing: ELISA ( optional gentyping), BDNF and COMT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm study: In this feasibility study, longitudinal mixed methods will be used to measure cognitive function and symptoms by objective tests, interviews, and biomarker assay in adults with brain cancer over time: prior to radiation (XRT; T1), 2-weeks post-XRT (T2), 2-3 months post-XRT (T3).
  Interventions: Other: Neuropsychological Testing

INTERVENTIONS:
Other: Neuropsychological Testing — Measure cognition function and cognitive reserve in patients before, during and after radiation therapy using cumulative scores of Hollingshead Index, North American Adult Reading Test, HVLT-R, TMT A&B and COWA over time.

SUMMARY:
Recent research indicates that variability in cognitive function for brain tumor survivors may be explained by differences in cognitive reserve (CR) and use of compensatory strategies.However, it is unknown when cognitive function declines or survivors tap into compensation. This longitudinal mixed methods study proposes to explore differences in cognitive function and change over time in newly diagnosed adults with brain cancer prior to, immediately after (within 2 weeks), and 2-3 months after radiation therapy treatment has been completed.

Specific aims are to:

Aim1: Examine the relationship between objective and subjective cognitive function in subjects newly diagnosed with brain cancer prior to and after XRT.

Aim 2: Explore the interrelationship between cognitive function and compensation (neural and behavioral) by high/low CR prior to and after XRT.

Aim 3: Describe the trajectory of objective and subjective cognitive function over time by CR, cancer type, and associated treatment-related factors.

DETAILED DESCRIPTION:
Cognitive impairments experienced by cancer survivors, from time of diagnosis through the health trajectory, are distressing, persistent, and negatively impact everyday function and quality of life. While reports of cancer- and treatment-related cognitive concerns vary substantially and may be underestimated in some diagnoses, the estimated incidence ranges from 30% in breast cancer up to 90% in brain cancers. Those with brain cancers, including both primary brain tumors and secondary brain metastases, often receive news of their diagnosis during prime productive years of their lives. Due to the cognitive effects from cancer or its treatment, most brain cancer survivors report difficulties returning to work or maintain family demands. Survivors often report co-occurring symptoms or a symptom cluster that include fatigue, sleep and mood disturbances, adding to multimorbidity conditions from the psychoneuroimmunologic effects of cancer. As medical advances have fostered significant gains in cancer survivorship and cancer is now recognized as a chronic illness, there is an urgency to address commonly faced symptoms and chronic conditions throughout the cancer trajectory beginning at time of diagnosis.

Cancer treatment is designed to induce cell death but when treating brain cancers, treatment may negatively impact neurogenesis and neural repair. Previous study indicates that some survivors of brain tumors use behavioral compensation, the investigators aim to understand how neural compensation may be impacted. Cognitive functions associated with biomarkers (NComp) are brain-derived neurotrophic factor (BDNF), catechol-O-methyl transferase (COMT). As survival rises, the investigators need to identify factors that moderate cognitive function in order to develop interventions aimed at minimizing functional decline.

This study is significant as it: 1) describes cognitive variability decline over time, and use of N/BComp; 2) uniquely explores cognition and N/BComp over time; 3) explores moderators of cognitive function across brain cancer survivors, 4) may lead to developing targeted cognitive interventions.

Cognitive function impacts everyday functional abilities and quality of life, however, change in cognition can elude detection. Discrepancies observed between subjective and objective cognitive, co-occurring symptoms, and its relationship with cognitive reserve are new research areas of interest in oncology. Exploring neural or behavioral compensation within the context of cognitive reserve is novel. No known oncology studies have reported the relationship of neural and behavioral compensation with change in cognitive function over time. Examining the trajectory of these variables can aid in identifying potential cognitive interventions for targeted use to prevent decline or maintain function over time.

This study is innovative because it is the first to explore the interface of neural/behavioral compensation and the cognitive trajectory, within a framework of cognitive reserve, in adults newly diagnosed with brain cancers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-65 years,
* Newly diagnosed with primary brain tumor or secondary brain metastases
* Able to read and write English as the neurocognitive testing will be administered using English language forms

Exclusion Criteria:

* Those with >moderate cognitive impairment (Mini-Mental Status Examination [MMSE] score<24) at baseline
* Aphasia
* Other neurodegenerative disorders Drink 3 or more alcoholic beverages per day (per Centers for Disease Control definition), report current use of illicit drugs/misuse of prescription medication, or currently undergoing treatment or had previous treatment for substance abuse at any time period (alcoholism or drug abuse).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the appropriate clinics within a large academic health care setting.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | Baseline, 2 weeks and 3 months post radiation therapy
  Serial neurocognitive testing using composite scores from the Trail Making A and B test
Change in cognitive function | Baseline, 2 weeks and 3 months post radiation therapy
  Serial neurocognitive testing using composite scores from the Controlled Oral Word Association (COWA) test
Change in cognitive function | Baseline, 2 weeks and 3 months post radiation therapy
  Serial neurocognitive testing using the composite scores from the Hopkins Verbal Learning Test

SECONDARY OUTCOMES:
Change in cognitive function | Baseline and up to 3 months post XRT
  Composite scores will be computed using the Functional Assessment of Cancer Cognition Scale
Change in cognitive function | Baseline and up to 3 months post XRT
  Composite scores will be computed using the Functional Assessment of Cancer-Treatment Cognition Scale
Change in cognition reserve | Baseline and up to 3 months post XRT
  Composite scores will be computed using the Hollingshead Index
Change in cognition reserve | Baseline and up to 3 months post XRT
  Composite scores will be computed using the North American Adult Reading Test

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Allen, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No